CLINICAL TRIAL: NCT01844999
Title: Personal Patient Profile - Prostate (P3P) II: Effectiveness-Implementation Trial in Diverse Health Care Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Donna Berry, PhD, RN, FAAN, ACON, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-363; 2R01NR009692-05 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Decision
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual patient education + standard educational websites (Other)
  Interventions: Behavioral: Standard prostate cancer information websites
- Usual patient education + P3P decision support website (Experimental)
  Interventions: Behavioral: Personal Patient Profile - Prostate (P3P)

INTERVENTIONS:
Behavioral: Personal Patient Profile - Prostate (P3P) — Website supporting informed patient decision making about prostate cancer care through tailored education and coaching
  Arms: Usual patient education + P3P decision support website
Behavioral: Standard prostate cancer information websites — Standard prostate cancer information websites (e.g., NCI, ASCO) presented to patients in addition to patient education that is usual in their clinics
  Arms: Usual patient education + standard educational websites

SUMMARY:
The purpose of this study is to determine whether using the P3P website can increase decisional preparation and satisfaction, and decrease decisional conflict, in men deciding how to manage early stage prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of prostate cancer, T1 or T2 of any risk level
* Biopsy done at enrolling site
* Upcoming appointment with consulting specialist at enrolling study site
* Able to read, write, understand English

Exclusion Criteria:

* Two or more post-biopsy specialist consults
* Begun treatment (or active surveillance)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | Change from baseline to 6-months
  O'Connor, 1995, Decisional conflict scale
Preparation for decision making | 1-month after study entry
  Graham and O'Connor, 1995, Preparation for decision making scale
Satisfaction with decision | 6-months after study entry
  Holmes-Rovner et al, 1996, Satisfaction with decision scale

SECONDARY OUTCOMES:
Concordance of care choice selected with self-reported influential personal preferences | 6-months from study entry
  Odds ratio of selecting a care option for prostate cancer concordant with avoiding prioritized side effects (XBRT or brachytherapy if concerned with sexual function; prostatectomy if concerned with bowel function; active surveillance if concerned with sexual, bowel, and/or bladder function; any treatment if not concerned with any side effect).
Net cost and benefit of the intervention | 1-week after study entry
  Cost to the patient will be measured in hours valued according to patient work status, income, and use of time. Benefit will be measured with Willingness to pay.
Time to treatment decision | 6-months from study entry
  Duration (in days) from pre-decision baseline questionnaire until patient decides on a care option for prostate cancer, either an active treatment type or active surveillance. Measured by patient recall at 6-months.

CONTACTS AND LOCATIONS:
Overall Officials: Donna L Berry, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Kaiser Permanente - Souther California, Downey, California
  - Kaiser Permanente - Southern California, Los Angeles, California
  - Emory Healthcare, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Pozzar RA, Xiong N, Hong F, Filson CP, Chang P, Halpenny B, Berry DL. Concordance between influential adverse treatment outcomes and localized prostate cancer treatment decisions. BMC Med Inform Decis Mak. 2022 Aug 24;22(1):223. doi: 10.1186/s12911-022-01972-w. PMID 36002847
- [Derived] Berry DL, Hong F, Blonquist TM, Halpenny B, Xiong N, Filson CP, Master VA, Sanda MG, Chang P, Chien GW, Jones RA, Krupski TL, Wolpin S, Wilson L, Hayes JH, Trinh QD, Sokoloff M. Decision regret, adverse outcomes, and treatment choice in men with localized prostate cancer: Results from a multi-site randomized trial. Urol Oncol. 2021 Aug;39(8):493.e9-493.e15. doi: 10.1016/j.urolonc.2020.11.038. Epub 2021 Jan 19. PMID 33353864
- [Derived] Wilson LS, Blonquist TM, Hong F, Halpenny B, Wolpin S, Chang P, Filson CP, Master VA, Sanda MG, Chien GW, Jones RA, Krupski TL, Berry DL. Assigning value to preparation for prostate cancer decision making: a willingness to pay analysis. BMC Med Inform Decis Mak. 2019 Jan 9;19(1):6. doi: 10.1186/s12911-018-0725-4. PMID 30626400